CLINICAL TRIAL: NCT01351103
Title: A Phase I, Open-label, Dose Escalation Study of Oral LGK974 in Patients With Malignancies Dependent on Wnt Ligands
Brief Title: A Study of LGK974 in Patients With Malignancies Dependent on Wnt Ligands
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLGK974X2101; 2011-000495-33 (EudraCT Number)
Record Dates: First submitted 2011-05-04; First posted 2011-05-10 (Estimated); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer; BRAF Mutant Colorectal Cancer; Melanoma; Triple Negative Breast Cancer; Head and Neck Squamous Cell Cancer; Cervical Squamous Cell Cancer; Esophageal Squamous Cell Cancer; Lung Squamous Cell Cancer
Keywords: LGK974; pancreatic adenocarcinoma; BRAF mutant colorectal cancer; RNF43 mutation; RSPO fusion; melanoma; triple negative breast cancer; PDR001; immunotherapy; head and neck scc; cervical scc; esophageal scc; lung scc
MeSH Terms: conditions — Pancreatic Neoplasms; Melanoma; Triple Negative Breast Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — LGK974; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LGK974 (Experimental): LGK974
  Interventions: Drug: LGK974
- LGK974 in combination with PDR001 (Experimental): LGK in combination with PDR001
  Interventions: Drug: LGK974; Biological: PDR001

INTERVENTIONS:
Drug: LGK974
  Other Names: WNT974
Biological: PDR001
  Arms: LGK974 in combination with PDR001

SUMMARY:
The primary purpose of this study was to find the recommended dose of LGK974 as a single agent and in combination with PDR001 that can be safely given to adult patients with selected solid malignancies that had progressed despite standard therapy or for which no effective standard therapy existed.

DETAILED DESCRIPTION:
This open-label multicenter phase 1 dose escalation study was the first to administer LGK974 as a single agent or in combination with PDR001 in humans.

The study comprised of 2 parts: a dose escalation of LGK974 as a single agent, followed by a safety expansion in specific disease indications; and a dose escalation of LGK974 in combination with PDR001, followed by a safety expansion in cutaneous melanoma.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of locally advanced or metastatic cancer that has progressed despite standard therapy or for which no effective standard therapy exists and histological confirmation of one of the following diseases indicated below:

Single Agent Dose escalation part:documented B-RAF mutant colorectal cancer or pancreatic adenocarcinoma. In addition, tumors of any histological origin with documented genetic alterations upstream in the Wnt signaling pathway are eligible with prior agreement with Novartis.

Single Agent Dose expansion part: documented B-RAF mutant colorectal cancer with documented RNF43 mutation and/or RSPO fusion or pancreatic adenocarcinoma with documented RNF43 mutation. In addition, patients with tumors of any histological origin with documented genetic alterations upstream in the Wnt signaling pathway (e.g. RNF43 or RSPO fusion) are eligible with prior agreement with Novartis

LGK974 with PDR001: Dose escalation: patients with the following cancers that were previously treated with anti-PD-1 therapy and whose best response on that therapy was progressive disease (i.e. primary refractory): melanoma, lung SCC, HNSCC. Patients with esophageal SCC, cervical SCC or TNBC who are either naïve or primary refractory to prior anti-PD-1 therapy.

LGK974 with PDR001: Dose expansion: patients with:

* cutaneous melanoma that was primary refractory to prior anti-PD-1 therapy, defined as a best response of progressive disease or stable disease for <= 4 months, or disease recurrence with the first 6 months of adjuvant therapy. Patients with BRAF V600-mutant melanoma must have also received and been failed by prior systemic therapy with BRAF V600 inhibitor, with or without a MEK inhibitor.
* Cutaneous melanoma with acquired resistance to prior anti-PD-1 therapy, defined as progressive disease following response (PR or CR) or following stable disease for > 4 months. Patients with BRAF V600-mutant melanoma must have also received and been failed by prior systemic therapy with a BRAF V600 inhibitor, with or without a MEK inhibitor.

Exclusion Criteria:

* Impaired cardiac function
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of LGK974 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection)
* Brain metastases that have not been adequately treated
* Malignant disease other than that being treated in this study
* Laboratory abnormalities as specified in the protocol
* Osteoporosis, osteopenia
* Bone fractures within the past year
* Pathologic bone fracture
* Active, known or suspected autoimmune disease or severe hypersensitivity reactions to other monoclonal antibodies

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) during the first cycle of LGK974 treatment and during the first 2 cycles of LGK974 in combination with PDR001 | 28 days (LGK974 single agent) and 56 days (LGK974 in combination with PDR001)
  DLT is defined as an adverse event or abnormal laboratory value that is assessed by the investigator as unrelated to disease, disease progression, intercurrent illness, or concomitant medications and that meets the criteria defined in the study protocol.
  The objective was to determine the Maximum Tolerated Dose (MTD) or Recommended Dose for Expansion (RDE) of LGK974 as a single agent and in combination with PDR001 when administered orally to adult patients with malignancies dependent on Wnt ligands.

SECONDARY OUTCOMES:
Type and category of study drug related adverse events (AE) | 61 months
  The incidence of treatment-emergent adverse events (new or worsening from baseline) will be summarized by primary system organ class, severity based on the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, type of AE, relationship to study drug by dose group.
Absorption and plasma concentrations of LGK974 | 61 months
  Evaluate pharmacokinetic (PK) parameters such as AUClast, AUCtau, Cmax, the apparent elimination T1/2 and Racc for LGK974 and its pharmacologically metabolite.
PD related to the Wnt pathway | 61 months
  Assessing percent change from baseline to post-treatment of PD related to the Wnt pathway.
Overall response rate of tumor | 61 months
  Patients with an Overall Response Rate(ORR), complete response (CR) or partial response (PR) rate and duration of response (DOR) assessed by RECIST 1.1 for single agent LGK974 and by RECIST1.1 and irRC for LGK974+PDR001.
Absorportion and plasma concentrations of PDR001 | 61 months
  Evaluate pharmacokinetic (PK) parameters such as AUClast, AUCtau, Cmax, the apparent elimination T1/2 and Racc for LGK974, its pharmacologically metabolite and PDR001.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- United States (6):
  - UCLA School of Medicine, Los Angeles, California
  - Sidney Kimmel Comprehensive Cancer Center Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute SC-7, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Onc Dept., Ann Arbor, Michigan
  - Karmanos Cancer Institute Wayne St, Detroit, Michigan
  - University of Texas/MD Anderson Cancer Center MD Anderson 2, Houston, Texas
- Novartis Investigative Site, Montreal, Quebec, Canada
- Novartis Investigative Site, Villejuif, France
- Novartis Investigative Site, Essen, Germany
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Napoli
- Netherlands (2):
  - Novartis Investigative Site, Rotterdam, South Holland
  - Novartis Investigative Site, Utrecht
- Spain (4):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodon J, Argiles G, Connolly RM, Vaishampayan U, de Jonge M, Garralda E, Giannakis M, Smith DC, Dobson JR, McLaughlin ME, Seroutou A, Ji Y, Morawiak J, Moody SE, Janku F. Phase 1 study of single-agent WNT974, a first-in-class Porcupine inhibitor, in patients with advanced solid tumours. Br J Cancer. 2021 Jul;125(1):28-37. doi: 10.1038/s41416-021-01389-8. Epub 2021 May 3. PMID 33941878
- See also: Link to Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18313